CLINICAL TRIAL: NCT01690260
Title: Bone Morphogenetic Protein-2 Increase as Substitute for Autologous Bone Graft After Ilizarow Treatment for Arthritis and Degenerative Bones.
Brief Title: Parallel Study Between BMP-2 and Autologous Bone Graft After Ilizarow Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Collaborators: Medtronic (Industry); Center for Clinical and Basic Research (CCBR A/S). (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N-20040019
Record Dates: First submitted 2012-09-12; First posted 2012-09-21 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Bone Degenerative Changes; Osteoarthritis; Degenerative Disorder of Bone
Keywords: Bone; Morphogenetic; Protein; Ilizarow; Autologous; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Bone Morphogenetic Protein 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bone Morphogenetic Protein 2 (Experimental): Condition of bone healing will be evaluated at serial radiological examinations and by clinical results according to a standard score system.
  Interventions: Drug: Bone Morphogenetic Protein 2; Procedure: Autologous bone graft
- Autologous bone graft (Experimental): Condition of bone healing will be evaluated at serial radiological examinations after 1,2,3,4,5,6,9 and 12 months. Blood tests and urine samples will also be examined for monitoring the bone healing process.
  Interventions: Drug: Bone Morphogenetic Protein 2; Procedure: Autologous bone graft

INTERVENTIONS:
Drug: Bone Morphogenetic Protein 2 — 12 mg recombinant BMP-2 combined with an injection of 1-2 g collagen type 1.
  Other Names: No other names.
Procedure: Autologous bone graft — Autologous bone graft in connection with bone docking operation.
  Other Names: No other names.

SUMMARY:
Results of growth factors indicate that Bone Morphogenetic Proteins (BMP) have an exceptional ability to stimulate different characteristics of mesenchymale cells to osseous cells. Local application of BMP results in an increase of osseous tissue regardless of the location of the growth factor.

5 years clinical studies show that BMP's can stimulate an increase of osseous tissue and improve clinical results when autologous bone graft is reduced or removed.

The purpose of this study is to examine whether recombinant growth factor BMP-2 can replace autologous bone graft in order to stimulating ossification during transplantation of osseous tissue.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalised for autologous bone graft based on Ilizarow treatment.
* Age between 20 and 70 years.

Exclusion Criteria:

* Rheumatoid osteoarthritis
* Malignant disease
* Current hormone treatment (glucocorticoid, parathyreoidea, thyreoidea)
* Pregnancy
* Abuse of drugs and alcohol
* Need of long-term NSAID treatment
* Breastfeeding women

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2004-09 (Actual); Primary Completion 2017-10-02 (Actual); Study Completion 2017-10-02 (Actual)

PRIMARY OUTCOMES:
Visible radiological signs of healing after 6 months. | An expected average of 6 months
  Radiological signs of healing is a criteria for a successful result.
  Failure of healing after 6 months and/or a need for stimulant bone healing intervention can result in:
  * Dynamic measurement af immobilization
  * Ultrasound stimulation
  * Re-surgery with application of bone graft or bone replacement

SECONDARY OUTCOMES:
Change in serologic bone markers | An expected average of 6 months
  Blood tests will be analyzed 1,2,3,4,6,9 and 12 months after operation in order to registrating a change in serologic bone markers.

CONTACTS AND LOCATIONS:
Overall Officials: Knud S. Christensen, MD, Principal Investigator — Orthopaedic Surgery Research Unit, Aalborg University Hospital, Denmark; David Donnell, Advisor, Study Chair — Medtronic Inc., Watford; Hans H. Hoeck, MD, Ph.D., Study Chair — Center for Clinical and Basic Research, Aalborg, Denmark (CCBR A/S)
Locations (1):
- Orthopaedic Surgery Research Unit, Aalborg University Hospital, Aalborg, Denmark